CLINICAL TRIAL: NCT06409832
Title: RimegepAnt effectIvenesS and tolErability as Migraine Preventive Treatment: a Prospective, Multicentric, Cohort Study (RAISE)
Brief Title: RimegepAnt effectIvenesS and tolErability as Migraine Preventive Treatment
Acronym: RAISE
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Società Italiana per lo Studio delle Cefalee (Other); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Università degli Studi dell'Aquila (Other); University of Roma La Sapienza (Other); Azienda Ospedaliero Universitaria Policlinico Modena (Other); Ospedale di Piove di Sacco (Unknown); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); A.O.U. Città della Salute e della Scienza (Other); Cliniche Humanitas Gavazzeni (Other); University of Campania Luigi Vanvitelli (Other); Ospedale Santo Stefano (Other); Azienda Policlinico Umberto I (Other); Auxologico San Luca (Other); Asst Degli Spedali Civili Di Brescia (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Luigi Francesco Iannone, Researcher at the Headache Center and Clinical Pharmacology Unit and the Department of Health Sciences, University of Florence, Principal Investigator, University of Florence
Other Study IDs: RICe_3
Record Dates: First submitted 2024-04-05; First posted 2024-05-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura; Chronic Migraine
Keywords: Headache; Medication overuse headache; Pain; Migraine prevention; Gepant; Rimegepant
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache; Headache Disorders, Secondary; Pain | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic migraine: Patients affected by an episodic pattern migraine(< 15 monthly headache days) with or without aura according to ICHD-III criteria.
  Interventions: Drug: Rimegepant 75 mg
- Chronic migraine: Patients affected by chronic migraine (> 15 monthly headache days with at least 8 days with migraine features) according to ICHD-III criteria.
  Interventions: Drug: Rimegepant 75 mg

INTERVENTIONS:
Drug: Rimegepant 75 mg — Patients using Rimegepant 75 mg orally disintegrating tablet every other day as migraine prevention
  Other Names: Rimegepant

SUMMARY:
The purpose of this prospective and multicentric study is to evaluate the effectiveness and tolerability of rimegepant as preventive migraine treatment in a cohort of episodic or chronic migraine patients.

DETAILED DESCRIPTION:
Rimegepant belongs to the gepants family, small molecules calcitonin gene- related peptide (CGRP) receptor antagonists. It is a new generation gepant, currently available as an orally disintegrating tablet at a single dose of 75 mg.

It has a double indication both for acute treatment for migraine with and without aura and preventive treatment of migraine. A previous randomized, placebo-controlled phase 2/3 trial demonstrated its effectiveness and tolerability in the preventive setting for patients with episodic and chronic migraine. Previous studies also demonstrated a good tolerability profile. The most commonly reported adverse events were nausea, nasopharyngitis, upper respiratory tract infections and urinary tract infections.

In this prospective multicentric study the investigators aim to evaluate rimegepant effectiveness and tolerability as preventive migraine treatment in a real-world setting. Subjects who meet the inclusion criteria will be enrolled and will participate in the study. Baseline demographic and clinical data will be collected at the baseline visit. The observation period will last for two years during which patients will take rimegepant 75 mg orally disintegrating tablet every other day for a time period related to eventual approval of reimbursability criteria.

Data will be collected at baseline and every three months for two years. Subjects will be asked to keep a headache diary to collect monthly headache and migraine days, migraine severity, associated symptoms and drug consumption. Questionnaires will be collected every three months.

Data collection will focus on: i) demographic data, ii) migraine history, iii) pain intensity, iv) presence and evolution of migraine associated symptoms and aura, v) migraine associated disability, vi) tolerability and eventual treatment- emergent adverse events, vii) treatment persistence, viii) questionnaires related to disability, allodynia, quality of life, interictal burden and effectiveness of the ongoing acute and preventive treatments. The online database REDCap will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the 3rd edition of the International Classification of Headache Disorder (ICHD-III);
* At least 4 monthly migraine days;
* Good compliance to study procedures;
* Availability of headache diary at least of the preceding months before enrollment.

Exclusion Criteria:

* Subjects with contraindications for use of gepants;
* Concomitant diagnosis of medical diseases and/or comorbidities that, in the Investigator's opinion might interfere with study assessments;
* medical comorbidities that could interfere with study results;
* Pregnancy and breastfeeding.
* Changes in preventive treatments in the month before the first administration of rimegepant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric study on patients attending the outpatient clinic of Italian Headache centres who meet criteria for rimegepant use for migraine preventive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Changes in migraine frequency after three months of treatment | Baseline (T0) - 3 months of treatment with rimegepant (T3)
  Changes in monthly migraine days after three months of treatment with rimegepant compared to baseline (continuous variable)
Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after three months of treatment with rimegepant | Baseline (T0) - 3 months of treatment with rimegepant (T3)
  Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after three months of treatment with rimegepant

SECONDARY OUTCOMES:
Changes in migraine frequency across twelve months of rimegepant treatment | Baseline (T0) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Change of monthly migraine days after six and twelve months of treatment with rimegepant compared to baseline (continuous variable)
Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) across twelve months of treatment with rimegepant | Baseline (T0) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after six and twelve months of treatment with rimegepant
Evaluation of any adverse event (qualitative) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Type of any adverse events in patients receiving rimegepant during the observation period (categorical variable)
Evaluation of any adverse event (quantitative) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Percentage of reported adverse events in patients receiving rimegepant during the observation period (continuous variable)
Evaluation of serious adverse event | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Percentage of serious adverse events (namely those resulting in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect) in patients receiving rimegepant during the observation period (continuous variable)
Evaluation of adverse event leading to treatment discontinuation | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Percentage of adverse events leading to treatment discontinuation in patients receiving rimegepant during the observation period (continuous variable)
Consistency of treatment response | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Percentage of patients with a stable 50% response during rimegepant treatment ( from 3 to 12 months of treatment) (continuous variable)
Changes in migraine disability (MIDAS) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in MIgraine Disability ASsement questionnaire across rimegepant treatment (continuous variable, 0-270 scale, higher scores indicate higher disability: 0-5, little/no disability; 6-10, mild disability; 11-20, moderate disability; >20, severe disability)
Changes in migraine disability (HIT-6) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in Headache Impact Test-6 questionnaire across rimegepant treatment (continuous variable, 36-78 scale, higher scores indicates greater disability)
Changes in response to acute migraine treatment (m-TOQ) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in migraine Treatment Optimization Questionnaire across rimegepant treatment (continuous variable, 0-8 scale, higher score indicates higher acute therapy effectiveness)
Changes in allodynia across rimegepant treatment (ASC-12) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in Allodynia Symptoms Checklist-12 questionnaire across rimegepant treatment (continuous variable, 0-24 scale, higher score indicates more severe allodynia)
Changes in quality of life across rimegepant treatment (MSQ) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in Migraine Specific Quality of life questionnaire across rimegepant treatment (continuous variable, 0-100 scale, 100 indicates full functionality)
Changes in interictal burden across rimegepant treatment (MIBS-4) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in Migraine Interictal Burden Scale-4 questionnaire across rimegepant treatment (continuous variable, 0-4 scale, 0 indicates no interictal burden, 1-2 mild level of interictal burden, 3 moderate interictal burden, 4 severe interictal burden)
Percentage of patients with Medication overuse headache reverted during treatment | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Percentage of patients with a baseline diagnosis of MOH reverted after 3 - 6 and 12 months of rimegepant treatment (continuous variable)

OTHER OUTCOMES:
Changes in the number of monthly migraine days with aura (quantitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in the number of monthly migraine days with aura across rimegepant treatment (continuous variable, through headache diary assessment)
Variation of duration of aura (qualitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in duration of aura across rimegepant treatment (categorical variable - minutes, assessed through headache diary)
Variation of type of aura (qualitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in type of aura across rimegepant treatment (assessed through headache diary and anamnestic data collection)
MMDs reduction in patients Non-responders to mAbs | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Change of monthly migraine days across rimegepant treatment in those patients who did not respond to anti-CGRP mAbs (continuous variable)
Percentage of 50% Responders in patients Non-responders to anti CGRP mAbs | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Percentage of 50% Responders across rimegepant treatment in those patients who did not respond to anti-CGRP mAbs (continuous variable)
Menstrually-related migraine | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Change in the number of menstrually-related attacks (according to ICHD-3) across rimegepant treatment compared to baseline (continuous variable)
Change in self-reported effectiveness of rimegepant treatment | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Change in Patients Global Impression of Change (PGIC) questionnaire across treatment (continuous variable, scale 0-7, 1 very much improved, 2 much improved, 3 minimally improved, 4 no change, 5 minimally worse, 6 much worse, 7 very much worse)
Changes in migraine severity | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in migraine severity (continuous variable, 0-10 numerical rating scale, higher scores indicate higher severity)
Changes in migraine duration across treatment | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in migraine duration across treatment (continuous variable, hours, assessed through a paper diary)
Changes in duration of the most bothersome symptom(s) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in duration of the most bothersome symptom(s) (continuous variable, minutes, assessed through a paper diary)
Changes in severity of the most bothersome symptom(s) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in severity of the most bothersome symptom(s) (continuous variable: 0-10 numerical rating scale, higher scores indicate higher severity)
Changes in self-reported effectiveness of acute treatment | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with rimegepant
  Changes in self-reported effectiveness of usual acute treatment (Patients Global Impression of Change questionnaire across treatment: continuous variable, scale 0-7, 1 very much improved, 2 much improved, 3 minimally improved, 4 no change, 5 minimally worse, 6 much worse, 7 very much worse)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - SOD Centro Cefalee e Farmacologia Clinica, AOU Careggi, Florence
  - IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia

REFERENCES:
- [Background] Lipton RB, Croop R, Stock EG, Stock DA, Morris BA, Frost M, Dubowchik GM, Conway CM, Coric V, Goadsby PJ. Rimegepant, an Oral Calcitonin Gene-Related Peptide Receptor Antagonist, for Migraine. N Engl J Med. 2019 Jul 11;381(2):142-149. doi: 10.1056/NEJMoa1811090. PMID 31291516
- [Background] Croop R, Lipton RB, Kudrow D, Stock DA, Kamen L, Conway CM, Stock EG, Coric V, Goadsby PJ. Oral rimegepant for preventive treatment of migraine: a phase 2/3, randomised, double-blind, placebo-controlled trial. Lancet. 2021 Jan 2;397(10268):51-60. doi: 10.1016/S0140-6736(20)32544-7. Epub 2020 Dec 15. PMID 33338437